CLINICAL TRIAL: NCT06973187
Title: A Phase 3, Open-Label, Randomized Study to Evaluate the Safety and Efficacy of BGB-16673 Compared to Pirtobrutinib in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: A Study to Evaluate the Safety and Efficacy of BGB-16673 Compared to Pirtobrutinib in Adults With Relapsed/Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-304; 2025-522860-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Noncovalent Bruton tyrosine kinase inhibitor; Bruton tyrosine kinase-targeted protein degrader
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: BGB-16673 (Experimental): Participants will receive BGB-16673 orally.
  Interventions: Drug: BGB-16673
- Arm B: Pirtobrutinib (Active Comparator): Participants will receive pirtobrutinib orally.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: BGB-16673 — BGB-16673 will be administered orally
  Arms: Arm A: BGB-16673
Drug: Pirtobrutinib — Pirtobrutinib will be administered orally
  Other Names: Jaypirca
  Arms: Arm B: Pirtobrutinib

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BGB-16673 alone compared with pirtobrutinib in patients with relapsed or refractory (R/R) chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) who had been previously treated with a covalent Bruton tyrosine kinase inhibitor (cBTKi).

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CLL or SLL, requiring treatment, based on 2018 iwCLL criteria
* Previously received treatment for CLL/SLL with a covalent Bruton tyrosine kinase inhibitor (cBTKi). Patients should have disease relapsed after or refractory to at least 1 line of therapy including a cBTKi.
* Participants with SLL must have measurable disease by computed tomography/magnetic resonance imaging, defined as ≥ 1 lymph node > 1.5 cm in longest diameter and measurable in 2 perpendicular diameters.

Exclusion Criteria:

* Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation.
* History of known bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
* History of ischemic stroke or intracranial hemorrhage within 6 months before first dose of study drug
* Prior exposure to any Bruton tyrosine kinase (BTK) protein degraders or noncovalent Bruton tyrosine kinase inhibitor (ncBTKi).
* Current or history of central nervous system involvement including the brain, spinal cord, leptomeninges, and cerebrospinal fluid (as documented by imaging, cytology, or biopsy) by CLL/SLL

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-04 (Actual); Primary Completion 2028-04-17 (Estimated); Study Completion 2028-04-17 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) per Independent Review Committee (IRC) | Up to approximately 3 years
  PFS is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by IRC using modified 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants with chronic lymphocytic leukemia (CLL) and Lugano classification for participants with small lymphocytic lymphoma (SLL).

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from the date of randomization to the date of death due to any cause.
PFS per Investigator (INV) | Up to approximately 3 years
  PFS per INV is defined as time from the date of randomization to the date of first disease progression or death, whichever occurs first, as determined by investigator using modified 2018 International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria for participants with CLL and Lugano classification for participants with SLL.
Overall Response Rate (ORR) per IRC and INV | Up to approximately 3 years
  ORR is defined as the percentage of participants with a best overall response of complete response, complete response with incomplete bone marrow recovery, nodular partial remission, or partial response, as assessed by the investigator and IRC using modified 2018 iwCLL criteria for patients with CLL and Lugano classification for patients with SLL.
Rate of Partial Response with Lymphocytosis (PR-L) or Higher per IRC and INV | Up to approximately 3 years
  The rate of PR-L or higher is defined as the percentage of participants with a best overall response of complete response, complete response with incomplete bone marrow recovery, nodular partial remission, partial response, or PR-L.
Duration of Response (DOR) per IRC and INV | Up to approximately 3 years
  DOR is defined as the time from initial response to disease progression or death, whichever occurs first.
Time to Next Anti-CLL/SLL Treatment (TTNT) | Up to approximately 3 years
  TTNT is defined as the time from the date of randomization to the date of next anti-CLL/SLL treatment.
Number of Participants with Adverse Events (AEs) | Up to approximately 3 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory abnormalities.
Change from Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire EORTC IL409 | Baseline and up to approximately 3 years
  EORTC IL409 consists of a set of 19 questions derived from the EORTC quality of life questionnaire core 30 (QLQ-C30) and its CLL module CLL17. The EORTC IL409 includes questions on global health status (GHS)/quality of life, physical functioning, role functioning, physical condition/fatigue, and symptom burden.Higher scores in GHS and functional scales and lower scores in symptom scales indicate better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (91):
- United States (23):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Stanford Cancer Institute, Palo Alto, California
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Titan Health Partners Llc Dba Astera Cancer Care, East Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Levine Cancer Institute (Lci), Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Dayton Physician Network, Dayton, Ohio
  - Tennessee Oncology, Pllc Nashville, Nashville, Tennessee
  - Blue Ridge Cancer Care (Oncology and Hematology Associates of Southwest Virginia), Roanoke, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Summit Cancer Centers, Spokane, Washington
  - Northwest Medical Specialties, Tacoma, Washington
  - Gunderson Health System, La Crosse, Wisconsin
- Australia (10):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Sunshine Coast Hospital and Health Service, Birtinya, Queensland
  - Flinders Medical Centre, Bedford PK, South Australia
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - Cabrini Hospital Malvern, Malvern East, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Medizinische Universitatsklinik Innsbruck, Innsbruck, Austria
- Belgium (3):
  - UZ GENT, Ghent
  - Az Groeninge Campus Loofstraat, Kortrijk
  - Chu Ucl Namur, Yvoir
- Hcfmusp Hospital Das Clinicas Da Faculdade de Medicina Da Universidade de Sao Paulo, São Paulo, Brazil
- France (8):
  - Centre de Lutte Contre Le Cancer Institut Bergonie, Bordeaux
  - Hopital Estaing, Clermontferrand
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital Saint Louis, Paris
  - Centre Henri Becquerel, Rouen
  - Iuc Toulouse Oncopole, Toulouse
  - Chu Tours Hopital Bretonneau, Tours
  - Chu Nancy Hopital Brabois, VandoeuvrelesNancy
- Gemeinschaftspraxis Fur Hamatologie Und Onkologie Dortmund, Dortmund, Germany
- Israel (6):
  - Bnai Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Meir Medical Center, KfarSava
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Di Padova, Padua
- Japan (8):
  - Matsuyama Red Cross Hospital, Matsuyama, Ehime
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hiroshima Red Cross Hospital and Atomic Bomb Survivors Hospital, Hiroshima, Hiroshima
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Kindai University Hospital, Sakai, Osaka
  - Cancer Institute Hospital of Jfcr, Kotoku, Tokyo
  - National Hospital Organization (Nho) Disaster Medical Center, Tachikawashi, Tokyo
  - Osaka Metropolitan University Hospital, Osaka
- New Zealand (3):
  - North Shore Hospital, Auckland
  - Tauranga Hospital, Tauranga
  - Wellington Regional Hospital (Ccdhb), Wellington
- Poland (5):
  - Copernicus Podmiot Leczniczy Sp Z Oo Wojewodzkie Centrum Onkologii, Gdansk
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej W Kielcach, Kielce
  - Szpital Kliniczny Mswia Z Warmisko Mazurskim Centrum Onkologii, Olsztyn
  - Narodowy Instytut Onkologii Im Marii Sklodowskiej Curie Hematology Unit, Warsaw
  - Uniwersytecki Szpital Kliniczny Im Jana Mikulicza Radeckiego We Wroclawiu, Wroclaw
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Romania (3):
  - Coltea Clinical Hospital, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj Napoca, ClujNapoca
  - Institutul Regional de Oncologie Iasi, Iași
- Singapore (2):
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital Haematology, Singapore
- South Korea (6):
  - Pusan National University Hospital, Seogu, Busan Gwang'yeogsi
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - The Catholic University of Korea, Seoul St Marys Hospital, SeochoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
- Spain (7):
  - Ico Badalona, Badalona
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario de Gran Canaria Dr Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen Del Rocio, Seville
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/